CLINICAL TRIAL: NCT03021226
Title: An Impact Evaluation of the Brothers United Fatherhood Program, a Community-Based Responsible Fatherhood Initiative
Brief Title: Evaluation of the Brothers United Fatherhood Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Economic Opportunity Planning Association dba Pathway, Inc. (Other)
Responsible Party: Principal Investigator, Michael Young, Ph.D., Principal Investigator, Economic Opportunity Planning Association dba Pathway, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90FK087-01-01
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Health Behavior
Keywords: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I: Adults (Experimental): Participants in Group I will be adults ages 20 to 24 years of age, 50 hours of instruction provided over a six-week period, and address three major topic areas: Fatherhood Development, Relationship Enhancement, and Financial Literacy/Work.
  Interventions: Behavioral: Fatherhood Development; Behavioral: Relationship Enhancement; Behavioral: Financial Literacy
- Group II: No Intervention: Adults (No Intervention): Participants in Group II will be adults ages 20 to 24 years of age who do not receive any hours of intervention.

INTERVENTIONS:
Behavioral: Fatherhood Development — Fatherhood Development is a curriculum based program provided by a facilitator through a skill-based education intervention.
  Arms: Group I: Adults
Behavioral: Relationship Enhancement — Relationship Enhancement is a curriculum based program provided by a facilitator through a skill-based education intervention.
  Arms: Group I: Adults
Behavioral: Financial Literacy — Relationship Enhancement is a curriculum based program provided by a facilitator through skill-based education intervention.
  Arms: Group I: Adults

SUMMARY:
The Brothers United Fatherhood Program (BUFP) will be conducting an evaluation that builds on literature and existing research from the healthy marriage/responsible fatherhood initiatives developed by ACF over the last 10 years, in particular the Supporting Healthy Marriage Program initiative that established a randomized clinical trial. The Brothers United Fatherhood Program will provide important data to expand the area of fatherhood development with the target population. This program is funded through an initiative of the Administration for Children and Families, Office of Family Assistance (OFA).

The study is intended to measure if the identified interventions improve the well-being and relationship between targeted participants and their families. The study intends to focus on the following outcomes:

* Demonstrate increased intake & knowledge of systems that help fathers
* Improvement in knowledge of employment & learn new opportunities for economic mobility
* Improvement communication & empathy skills towards partner
* Increase in understanding of healthy marriage & its value to fathers
* Demonstrate an understanding of financial planning
* Demonstrate improved conflict resolution, behavior patterns, including those leading to domestic violence
* Increase in reports of improved adult & child relationships
* Demonstrate an increase job readiness skills such as employment preparedness & career direction

DETAILED DESCRIPTION:
Do those who participate in the program result in more positive self-reported attitudes and behaviors than the control group relative to the following:

1. Improved healthy relationship and marriage skills.
2. Improved co-parenting skills
3. Increased frequency of father/child engagement
4. Increased financial responsibility of fathers
5. Progress toward a greater economic stability, including skill attainment and employment.
6. Reduce recidivism?

This reflects intention-to-treat (ITT) analysis where all participants who are enrolled and randomly assigned to treatment are included in the analysis regardless of their adherence with the entry criteria, regardless of subsequent withdrawal from treatment or deviation from the protocol. This will preserve the pragmatic balance generated by the original random treatment allocation.

Also, "per protocol analysis" will be conducted to evaluate if full project participation results in more positive self-reported attitudes and behaviors than the control group participants.

What personal characteristics and other external factors are related to achieving successful outcomes in the program?

ELIGIBILITY:
Inclusion Criteria:

* Participants must be parents between the ages of 20 to 24.

Exclusion Criteria:

* Participants cannot be younger than 20 years of age.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Fatherhood Development measured with a Questionnaire | At program enrollment-during registration, immediately after completing intervention, and at 1 year follow up.
  Fatherhood Development - Questionnaire developed for intervention to measure change from before intervention to immediately after intervention, and at 1 year after completion.

SECONDARY OUTCOMES:
Relationship Enhancement measured with a Questionnaire | At program enrollment-during registration, immediately after completing intervention, and at 1 year follow up.
  Relationship Enhancement - Questionnaire developed for intervention to measure change from before intervention to immediately after intervention, and at 1 year after completion.
Financial Literacy/Work Skills measured with a Questionnaire | At program enrollment-during registration, immediately after completing intervention, and at 1 year follow up.
  Financial Literacy/Work Skills - Questionnaire developed for intervention to measure change from before intervention to immediately after intervention, and at 1 year after completion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Young, PHD, Principal Investigator — Center for Evidence-Based Programming
Locations (1):
- Pathway, Inc., Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No